CLINICAL TRIAL: NCT00860574
Title: A Multi-Center Study of Conditioning With Treosulfan, Fludarabine and Escalating Doses of TBI for Allogeneic Hematopoietic Cell Transplantation in Patients With Acute Myeloid Leukemia (AML) Myelodysplastic Syndrome (MDS), and Acute Lymphoblastic Leukemia (ALL)
Brief Title: Treosulfan, Fludarabine Phosphate, and Total-Body Irradiation Before Donor Stem Cell Transplant in Treating Patients With High-Risk Acute Myeloid Leukemia, Myelodysplastic Syndrome, Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Joachim Deeg, Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2272.00; NCI-2010-00315 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P01HL036444 (NIH)
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-02

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Blastic Phase Chronic Myelogenous Leukemia; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Chronic Myelogenous Leukemia; Childhood Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — treosulfan; fludarabine phosphate; Whole-Body Irradiation; Peripheral Blood Stem Cell Transplantation; Tacrolimus; Transplantation; Methotrexate; merphos

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (allogeneic transplantation) (Experimental): CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV over 30 minutes on days -6 to day -2 and treosulfan IV over 2 hours on days -6 to day -4. Patients also undergo total-body irradiation on day 0. TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplantation or bone marrow transplantation on day 0. GVHD PROPHYLAXIS: Patients receive tacrolimus IV continuously or PO BID on days -1 to 56, followed by a taper until day 180 in the absence of GVHD. Patients also receive methotrexate IV on days 1, 3, 6, and 11.
  Interventions: Drug: treosulfan; Drug: fludarabine phosphate; Radiation: total-body irradiation; Procedure: peripheral blood stem cell transplantation; Drug: tacrolimus; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Drug: methotrexate

INTERVENTIONS:
Drug: treosulfan — Given IV
  Other Names: dihydroxybusulfan; Ovastat; tresulfon
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Radiation: total-body irradiation — Low dose starting at 2Gy
  Other Names: TBI
Procedure: peripheral blood stem cell transplantation — Given IV per institutional standard practice
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Drug: tacrolimus — Given IV or PO
  Other Names: FK 506; Prograf
Procedure: allogeneic bone marrow transplantation — Given IV per institutional standard practice
  Other Names: bone marrow therapy, allogeneic; bone marrow therapy, allogenic; transplantation, allogeneic bone marrow; transplantation, allogenic bone marrow
Procedure: allogeneic hematopoietic stem cell transplantation — Given IV per institutional standard practice
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX

SUMMARY:
This phase II trial is studying how well giving treosulfan together with fludarabine phosphate and total-body irradiation followed by donor stem cell transplant works in treating patients with high-risk acute myeloid leukemia, myelodysplastic syndrome, acute lymphoblastic leukemia. Giving chemotherapy, such as treosulfan and fludarabine phosphate, and total-body irradiation before a donor bone marrow or peripheral blood stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving tacrolimus and methotrexate before and after transplant may stop this from happening

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Decrease the incidence of relapse to < 15% at 6 month post transplant in patients with high risk acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) transplanted from related or unrelated donors, without unacceptably increasing toxicity (10% non-relapse mortality [NRM] at 6 months).

SECONDARY OBJECTIVES:

I. Evaluate the incidence of NRM at 180 days and 1 year after hematopoietic cell transplantation (HCT).

II. Evaluate overall survival (OS) and relapse-free survival (RFS). III. Incidence of grades II-IV acute graft-versus-host disease (GVHD). IV. Incidence of chronic GVHD. V. Donor chimerism on days +28 and +100.

OUTLINE:

CONDITIONING REGIMEN: Patients receive fludarabine phosphate intravenously (IV) over 30 minutes on days -6 to day -2 and treosulfan IV over 2 hours on days -6 to day -4. Patients also undergo total-body irradiation on day 0.

TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplantation or bone marrow transplantation on day 0.

GVHD PROPHYLAXIS: Patients receive tacrolimus IV continuously or orally (PO) twice daily (BID) on days -1 to 56, followed by a taper until day 180 in the absence of GVHD. Patients also receive methotrexate IV on days 1, 3, 6, and 11.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia (AML):

  * All AML patients beyond 1st remission;
  * Intermediate or high risk AML patients (based on South West Oncology Group [SWOG] cytogenetic criteria) in 1st complete remission
* Myelodysplastic syndrome (MDS)
* Other myeloid malignancies as chronic myelogenous leukemia (CML), CML accelerated phase, CML blast crisis, chronic myelomonocytic leukemia (CMML) (to be approved by patient care conference [PCC])
* With Karnofsky Index or Lansky Play-Performance Scale > 70% on pre-transplant evaluation
* Able to give informed consent (if > 18 years), or with a legal guardian capable of giving informed consent (if < 18 years)
* Previous autologous or allogeneic HCT is allowed
* Donors must be:

  * Human leukocyte antigen (HLA)-identical related donors or
  * Unrelated donors matched for HLA-A, B, C, DRB1, and DQB1 defined by high resolution deoxyribonucleic acid (DNA) typing or mismatched for one HLA allele, except for HLA-C where no mismatch is allowed
  * Able to undergo peripheral blood stem cell collection or bone marrow harvest
  * In good general health, with a Karnofsky or Lansky Play Performance score > 90%
  * Able to give informed consent (if > 18 years), or with a legal guardian capable of giving informed consent (if < 18 years)
* Acute lymphoblastic leukemia (ALL): all ALL patients not eligible for other protocols

Exclusion Criteria:

* Receiving umbilical cord blood
* With impaired cardiac function as evidenced by ejection fraction < 35% or cardiac insufficiency requiring treatment or symptomatic coronary artery disease
* With impaired pulmonary function as evidenced by partial pressure of oxygen (pO2) < 70 mm Hg and diffusing capacity of the lung for carbon monoxide (DLCO) < 70% of predicted or pO2 < 80 mm Hg and DLCO < 60% of predicted; or receiving supplementary continuous oxygen
* With impaired renal function as evidenced by creatinine-clearance < 50% for age, weight, height or serum creatinine > 2x upper normal limit or dialysis-dependent
* With hepatic dysfunction as evidenced by total bilirubin or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.0 x upper normal limit or evidence of synthetic dysfunction or severe cirrhosis
* With active infectious disease requiring deferral of conditioning, as recommended by an Infectious Disease specialist
* With human immunodeficiency virus (HIV)-positivity or active infectious hepatitis because of possible risk of lethal infection when treated with immunosuppressive therapy
* With central nervous system (CNS) leukemic involvement not clearing with intrathecal chemotherapy and/or cranial radiation prior to initiating conditioning (day -6)
* With life expectancy severely limited by diseases other than malignancy
* Women who are pregnant or lactating because of possible risk to the fetus or infant
* With known hypersensitivity to treosulfan and/or fludarabine
* Receiving another experimental drug within 4 weeks before initiation of conditioning (day -6)
* Unable to give informed consent (if > 18 years) or with a legal guardian (if < 18 years) unable to give informed consent
* Ineligible donors will be those:

  * Deemed unable to undergo marrow harvesting or PBSC mobilization and leukapheresis
  * Who are HIV-positive
  * With active infectious hepatitis
  * Females with a positive pregnancy test
  * Unable to give informed consent (if > 18 years) or with a legal guardian (if < 18 years) unable to give informed consent

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2009-02; Primary Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boglarka Gyurkocza, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - University of Colorado, Denver, Colorado
  - Oregon Health and Science University, Portland, Oregon
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Allogeneic Transplantation)
Started | 96
Completed | 93
Not Completed | 3
Not completed — Death | 2
Not completed — Relapse | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Allogeneic Transplantation): CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV over 30 minutes on days -6 to day -2 and treosulfan IV over 2 hours on days -6 to day -4. Patients also undergo total-body irradiation on day 0. TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplantation or bone marrow transplantation on day 0. GVHD PROPHYLAXIS: Patients receive tacrolimus IV continuously or PO BID on days -1 to 56, followed by a taper until day 180 in the absence of GVHD. Patients also receive methotrexate IV on days 1, 3, 6 and 11.
  treosulfan: Given IV
  fludarabine phosphate: Given IV
  total-body irradiation: Low dose starting at 2Gy
  peripheral blood stem cell transplantation: Given IV per institutional standard practice
  tacrolimus: Given IV or PO
  allogeneic bone marrow transplantation: Given IV per institutional standard practice
  allogeneic hematopoietic stem cell transplantation: Given IV per institutional standard practice
  methotrexate: Given IV
Arm/Group | Treatment (Allogeneic Transplantation)
Number analyzed (Participants) | 96
Age, Continuous [Median (Full Range); unit: years] | 51 [1 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 93
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 1
  White | 87
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 96

OUTCOME MEASURES:

1. Primary Outcome: Relapse Incidence
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic Transplantation)
Number analyzed (Participants) | 96
Participants | 18

2. Primary Outcome: Non Relapse Mortality (NRM) Incidence
Description: Cumulative incidence of NRM at 6 months. NRM includes all deaths without relapse or disease progression.
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic Transplantation)
Number analyzed (Participants) | 96
Participants | 6

3. Secondary Outcome: Non Relapse Mortality Incidence
Time Frame: 1 year after HCT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic Transplantation)
Number analyzed (Participants) | 96
Participants | 6

4. Secondary Outcome: Overall Survival (OS)
Time Frame: at 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic Transplantation)
Number analyzed (Participants) | 96
Participants | 71

5. Secondary Outcome: Relapse-free Survival
Time Frame: at 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic Transplantation)
Number analyzed (Participants) | 96
Participants | 62

6. Secondary Outcome: Incidence of Grades II-IV Acute GVHD
Time Frame: at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic Transplantation)
Number analyzed (Participants) | 96
Participants | 57

7. Secondary Outcome: Incidence of Chronic GVHD
Time Frame: at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic Transplantation)
Number analyzed (Participants) | 96
Participants | 20

8. Secondary Outcome: Median Donor CD3 + T Lymphocyte Chimerism in Peripheral Blood
Description: Donor chimerism was evaluated in peripheral blood T cells
Time Frame: Day 28 after HCT
Measure: Median (Full Range); unit: percentage of T cells
Arm/Group | Treatment (Allogeneic Transplantation)
Number analyzed (Participants) | 87
percentage of T cells | 100 [88 to 100]

ADVERSE EVENTS:
Time Frame: Toxicities Before Day 100
Description: Toxicities documented per Common Terminology Criteria for Adverse Events (CTCAE) v3.0
Arm/Group | Treatment (Allogeneic Transplantation)
All-Cause Mortality (participants affected / at risk) | 21/96
Serious Adverse Events (participants affected / at risk) | 17/96
Other Adverse Events (participants affected / at risk) | 68/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Allogeneic Transplantation) (N=96)
Mucositis (Gastrointestinal disorders) | 4
Bacterial/sepsis (Infections and infestations) | 1
Heart failure (Cardiac disorders) | 1
Gut GVHD (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 4
VRE bacteremia/sepsis (Infections and infestations) | 1
Disseminated toxoplasmosis (Infections and infestations) | 1
Enterococcal bacteremia/VRE (Infections and infestations) | 1
CMV pneumonia (Infections and infestations) | 1
Aspirgillus (Infections and infestations) | 1
Hypotension (Cardiac disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Acute respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia/resp failure (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Intubated secondary to DAH (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure/intubated (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac arrythmia (Respiratory, thoracic and mediastinal disorders) | 1
Pul.Edema (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Bilirubin (Hepatobiliary disorders) | 1
Liver failure (Hepatobiliary disorders) | 1
AST 2680 (Hepatobiliary disorders) | 1
Hypoglycemia w/seizures (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Diffuse alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Kidney rejection - pre-existing hx kidney transplant (Renal and urinary disorders) | 1
Renal failure/dialysis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Apnea (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Allogeneic Transplantation) (N=96)
Mucositis (Gastrointestinal disorders) | 23
Mucosi (Gastrointestinal disorders) | 2
Infections (Infections and infestations) | 56
Deep vein thrombosis (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 6
Adrenal insufficiency (General disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6
Retinal central vein occlusion (Eye disorders) | 1
Dehydration (General disorders) | 2
Proximal myopathy (General disorders) | 1
Steroid induced DM (General disorders) | 1
LE weakness/deconditioning (General disorders) | 1
Fall (General disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 11
Diverticulitis (Gastrointestinal disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Other (Gastrointestinal disorders) | 1
Pain (Musculoskeletal and connective tissue disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 1
Neuropathic leg pain (Nervous system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 3
Edema (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 4
LVEF 35% (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 11
ALT/AST (Hepatobiliary disorders) | 1
ALT (Hepatobiliary disorders) | 1
AST (Hepatobiliary disorders) | 2
t.bili 4.2 (Hepatobiliary disorders) | 1
Bilirubin (Hepatobiliary disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Steroid myopathy (Musculoskeletal and connective tissue disorders) | 2
Elevated ferritin (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
GI bleed (Gastrointestinal disorders) | 1
Confusion (Psychiatric disorders) | 4
Altered Mental Status (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Acute renal failure/creatinine (Renal and urinary disorders) | 2
Creatinine (Renal and urinary disorders) | 1
Renal failure/acidosis (Renal and urinary disorders) | 1
Syncope (Nervous system disorders) | 2
Peripheral neuropathy (Nervous system disorders) | 1
Hallucinations (Psychiatric disorders) | 1
Posterior reversible encephalopathy syndrome (PRES) (Nervous system disorders) | 1
Malnutrition (General disorders) | 1
Thrombotic thrombocytopenic purpura (TTP) coagulation (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No